CLINICAL TRIAL: NCT03179046
Title: Association of Heart Structure and Function Abnormalities With Laboratory Findings in Patients With Systemic Lupus Erythematosus
Brief Title: Cardiac and Laboratory Findings in Patients With Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Assistant lecturer, Assiut University
Other Study IDs: 17200078
Record Dates: First submitted 2017-06-04; First posted 2017-06-07 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Laboratory tests and cardiac imaging — Laboratory tests (blood count, liver and kidney functions, antibodies, acute phase reactants), Echocardiography and gadolinium enhanced cardiac MRI

SUMMARY:
This study is designed to investigate the association of the clinical and laboratory parameters or data with the cardiac structural and functional abnormalities in systemic lupus erythematosus(SLE). Patients with at least four ACR classification criteria for SLE and stable clinical condition (no need for immunosuppressive therapy intensification, i.e. current immunosuppressive drug dose increase or introduction of an additional immunosuppressive drug within last 3 months) will be included in the study. Study procedures will include clinical evaluation, lab tests including blood counts, liver and kidney functions and antibodies levels such as ANA, antiphospholipid antibodies, anti-ds DNA as well as inflammatory markers such as sedimentation rates. Also evaluation of cardiac status by cardiologist examination echocardiography and gadolinium enhanced cardiac MRI. Next, correlation between cardiac abnormalities and laboratory changes will be statistically analyzed.

DETAILED DESCRIPTION:
* Subject recruitment and obtaining consent Study subjects (SLE patients) will be recruited from patients attending outpatient clinic and inpatients of the Rheumatology and Rehabilitation Department, Faculty of Medicine, Assiut University. Written informed consent form will be obtained from each patient.
* Baseline evaluation:

  1. All SLE patients selected for the study will fulfill the ACR criteria for the diagnosis of SLE .
  2. Thorough clinical history and examination will be performed to all SLE patients. Pulmonary function (PFTs) test will be performed to exclude respiratory failure.
  3. Urine pregnancy test to exclude pregnancy will be performed to all SLE females' patients of the childbearing period in the study group.
* Laboratory tests: the following tests will be performed to all study population:

  1. Complete blood count (CBC),
  2. Liver and kidney functions and measurement of protein in urine collected over 24 hours,
  3. Levels of Erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP).
  4. Antinuclear antibodies (ANA) and their titer will be assessed by indirect immunofluorescence,
  5. Complement system C3 and C4 factors will be measured to determine disease activity,
  6. Serum levels of anticardiolipin (aCL) and lupus anticoagulant antibodies will be measured using ELISA.
* Disease activity will be assessed by using SELDAI score [11].
* Cardiac evaluation

  1. Echocardiography will be performed to evaluate structural and functional outcome measures.
  2. Cardiac MRI: Multiple consecutive MR image sections will be obtained from the apex to the base of the heart. T2 and T1 mapping will be performed. T1-weighted inversion recovery scout images will be acquired 15 min after injection of 0.2 mmol/kg of gadolinium based contrast agent. The functional and volumetric analysis will be performed to quantify ventricular volumes and functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients have at least four ACR classification criteria for SLE.
* Stable clinical condition (no need for immunosuppressive therapy intensification, i.e. current immunosuppressive drug dose increase or introduction of an additional immunosuppressive drug within last 3 months).

Exclusion Criteria:

* Patients less than 18 years old
* Clinical symptoms of heart failure.
* Renal failure (creatinine clearance < 30 ml/ min).
* Respiratory failure.
* Pregnancy.
* Patients with contraindications for MRI e.g. patients with aneurysm clips or cardiac pacemakers and patients who are sensitive to gadolinium dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients have at least four ACR classification criteria for SLE.
  * Stable clinical condition (no need for immunosuppressive therapy intensification, i.e. current immunosuppressive drug dose increase or introduction of an additional immunosuppressive drug within last 3 months).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation between echocardiographic parameters and the presence of autoantibodies as well as the concentration of CRP and complement C3 and C4 components. | 1year
  Correlation between echocardiographic parameters (left ventricle diastolic and systolic dimensions, its ejection fraction, thickness of the walls in diastole, left atrium diameter, right ventricle diastolic diameter, ascending aorta diameter, mitral and tricuspid inflow velocity, valvular pressure gradients, regurgitation assessment , thickness of pericardium and the presence of pericardial effusion) and the presence of autoantibodies as well as the concentration of CRP and complement C3 and C4 components.
The presence of subclinical myocarditis, assessment of coronary blood flow, left and right ventricle as shown by cardiac MRI and its correlation with autoantibodies. | 1 year
  The presence of subclinical myocarditis, assessment of coronary blood flow, left and right ventricle (including ventricular size, thickness, wall motion, and ejection fraction) as shown by cardiac MRI(Multiple consecutive MR image sections will be obtained from the apex to the base of the heart. T2 and T1 mapping will be performed. T1-weighted inversion recovery scout images will be acquired 15 min after injection of 0.2 mmol/kg of gadolinium based contrast agent. The functional and volumetric analysis will be performed to quantify ventricular volumes and functions.
  ) and its correlation with autoantibodies.
Correlation between cardiac abnormalities (evaluated with Echocardiography and cardiac MRI) and disease activity evaluated with SELDAI score. | 1 year
  Correlation between cardiac abnormalities(evaluated with Echocardiography and cardiac MRI) and disease activity evaluated with SELDAI score.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Facultu of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No